CLINICAL TRIAL: NCT02232386
Title: A Phase 2 Multicenter Study to Assess the Activity and the Safety of Front-line Ibrutinib Plus Rituximab (IR) in Unfit Patients With Chronic Lymphocytic Leukemia (CLL).
Brief Title: Phase 2 Study to Assess Activity & Safety of Front-line Ibrutinib + Rituximab in Unfit Chronic Lymphocytic Leukemia
Acronym: LLC1114
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Gruppo Italiano Malattie EMatologiche dell'Adulto (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: LLC1114; 2014-002714-23 (EudraCT Number)
Record Dates: First submitted 2014-09-02; First posted 2014-09-05 (Estimated); Last update posted 2025-01-16 (Actual); Status verified 2025-01

CONDITIONS: Chronic Lymphocyte Leukemia; Adult Patients
Keywords: Chronic lymphocyte leukemia; Adults; Ibrutinib
MeSH Terms: interventions — ibrutinib; Rituximab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Treatment (Experimental): Ibrutinib (PCI-32765) 420 mg (3 x 140 mg capsules) will be administered orally once daily. The first dose will be delivered in the clinic on Day 1, after which subsequent dosing is typically on an outpatient basis. Treatment duration with Ibrutinib will be based on what comes first of the following three options:
  * Treatment until progression or toxicity
  * Treatment until MRD negativity for 6 months
  * Treatment for 6 years. Rituximab 375 mg/m2 iv. Month 1: day 1 of weeks 1, 2, 3, 4; months 2-6: day 1of week 1.
  Interventions: Drug: Ibrutinib; Drug: Rituximab

INTERVENTIONS:
Drug: Ibrutinib — Ibrutinib (PCI-32765) 420 mg (3 x 140 mg capsules) will be administered orally once daily. The first dose will be delivered in the clinic on Day 1, after which subsequent dosing is typically on an outpatient basis.
Drug: Rituximab — Rituximab 375 mg/m2 iv. Month 1: day 1 of weeks 1, 2, 3, 4; months 2-6: day 1of week 1.

SUMMARY:
The present study aims at evaluating whether treatment with two different drugs, Ibrutinib and Rituximab is both efficient and safe for newly diagnosed patients with chronic lymphocytic leukemia.

DETAILED DESCRIPTION:
Given that:

* Ibrutinib as single agent has been associated with a high response rate and PFS in previously treated patients, and in patients with poor prognosis clinical and biologic features.
* Ibrutinib as single agent has proven activity and is associated with a good safety profile in elderly patients with CLL.
* The Ibrutinib plus Rituximab combination has been associated with a high response rate and PFS in previously treated patients, and in patients with poor prognosis clinical and biologic features.
* The combined administration of Ibrutinib and Rituximab could be an effective and safe front-line treatment schedule for unfit patients with CLL.
* The current study is designed to evaluate whether first line treatment with Ibrutinib and Rituximab results in a significant improvement in PFS at 12 months as compared with chlorambucil plus rituximab in patients unfit for fludarabine- or bendamustine-based treatments.

ELIGIBILITY:
Inclusion Criteria:

1. 18 years of age or older.
2. Diagnosis of CLL meeting IWCLL criteria.
3. The diagnosis of CLL requires a history of lymphocytosis with a B-lymphocyte count ≥5,000/μL. Prolymphocytes may comprise no more than 55% of blood lymphocytes.
4. Active disease meeting at least 1 of the following IWCLL 2008 criteria for requiring treatment:

   1. Evidence of progressive marrow failure as manifested by the development of, or worsening of, anemia or thrombocytopenia.
   2. Massive (ie, at least 6 cm below the left costal margin), progressive, or symptomatic splenomegaly.
   3. Massive nodes (ie, at least 10 cm in longest diameter), progressive, or symptomatic lymphadenopathy.
   4. Progressive lymphocytosis with an increase of more than 50% over a 2-month period or a lymphocyte doubling time (LDT) of less than 6 months (which may be extrapolated). Lymphocyte doubling time can be obtained by linear regression extrapolation of ALCs obtained at intervals of 2 weeks over an observation period of 2 to 3 months. For patients with initial blood lymphocyte counts of less than 30 x 109/L (30,000/μL), LDT should not be used as a single parameter to define indication for treatment. In addition, factors contributing to lymphocytosis or lymphadenopathy other than CLL (eg, infections) should be excluded.
   5. Constitutional symptoms, defined as 1 or more of the following disease-related symptoms or signs:

      * Unintentional weight loss >10% within the previous 6 months prior to screening
      * Significant fatigue (inability to work or perform usual activities)
      * Fevers higher than 38.0°C for 2 or more weeks without evidence of infection; or
      * Night sweats for more than 1 month without evidence of infection
      * Measurable nodal disease by computed tomography (CT). Measurable nodal disease is defined as at least one lymph node >1.5 cm in longest diameter in a site that has not been previously irradiated. An irradiated lesion may be assessed for measurable disease only if there has been documented progression in that lesion since radiotherapy has ended.
5. No prior treatment.
6. Total CIRS >6 and/or creatinine clearance <70 ml/min [Cockcroft-Gault]).
7. Hematology values within the following limits: Absolute neutrophil count (ANC) ≥1 x 109/L (ie, ≥1000/μL) independent of growth factor support. Platelets ≥50,000/mm3 if bone marrow involvement independent of transfusion support
8. Biochemical values within the following limits:

   1. Alanine aminotransferase (ALT) and aspartate aminotransferase (AST) ≤3 x upper limit of normal (ULN)
   2. Total bilirubin ≤1.5 x ULN unless bilirubin rise is due to Gilbert's syndrome or of non-hepatic origin
   3. Serum creatinine ≤2 x ULN or estimated Glomerular Filtration Rate (Cockroft Gault) ≥40 mL/min
9. Women of childbearing potential and men who are sexually active must be practicing a highly effective method of birth control during and after the study consistent with local regulations regarding the use of birth control methods for subjects participating in clinical trials. Men must agree not to donate sperm during and after the study. For females, these restrictions apply for 1 month after the last dose of study drug. For males, these restrictions apply for 3 months after the last dose of study drug.
10. Women of childbearing potential must have a negative serum (beta-human chorionic gonadotropin [β-hCG]) or urine pregnancy test at Screening. Women who are pregnant or breastfeeding are ineligible for this study.
11. A signed (or signed by their legally-acceptable representatives) informed consent document indicating that they understand the purpose of and procedures required for the study, including biomarkers, and are willing to participate in the study.

Exclusion Criteria:

1. Any significant concurrent, uncontrolled medical condition or organ system dysfunction and/or laboratory abnormality or psychiatric disease which, in the investigator's opinion, could compromise the subject's safety, interfere with the absorption or metabolism of ibrutinib capsules, or put the study outcomes at undue risk or prevent the subject from signing the informed consent form.
2. Pregnant or lactating females
3. Known presence of alcohol and/or drug abuse.
4. Any potential subject who meets any of the following criteria will be excluded from participating in the study.
5. Major surgery within 4weeks of randomization.
6. Uncontrolled autoimmune hemolytic anemia or thrombocytopenia.
7. Known central nervous system lymphoma.
8. History of stroke or intracranial hemorrhage within 6 months prior to randomization, or of a significant cerebrovascular disease in the past 6 months or ongoing event with active symptoms or sequelae.
9. Requires anticoagulation with warfarin or equivalent vitamin K antagonists (eg, phenprocoumon) in any moment of the study.
10. Requires treatment with strong CYP3A inhibitors.
11. Clinically significant cardiovascular disease such as uncontrolled or symptomatic arrhythmias, congestive heart failure, or myocardial infarction within 6 months of Screening, or any Class 3 (moderate) or Class 4 (severe) cardiac disease as defined by the New York Heart Association
12. Vaccinated with live, attenuated vaccines within 4 weeks of randomization.
13. Known history of human immunodeficiency virus (HIV) positive serology for HIV; active Hepatitis B Virus infection or positive serology for Hepatitis B (HBV) defined as a positive test for HBsAg and HBV-DNA; active Hepatitis C or HCV-RNA positive; any uncontrolled active systemic infection requiring intravenous (IV) antibiotics, antifungal, or antiviral treatment such as, but not limited to, chronic renal infection, chronic chest infection; history of tuberculosis within the last five years or recent exposure to tuberculosis equal to or less than 6 months.
14. Richter's syndrome (RS), concomitant or past malignancy. Subjects who have been free of malignancy for at least 5 years, or have a history of completely resected non-melanoma skin cancer, or successfully treated in situ carcinoma are eligible.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 156 (Actual)
Dates: Start 2015-03-02 (Actual); Primary Completion 2018-04 (Actual); Study Completion 2024-04-16 (Actual)

PRIMARY OUTCOMES:
Number of patients on progression-free survival | At 12 months from treatment start
  To estimate Progression-Free Survival (PFS) at 12 months in patients treated with Ibrutinib plus Rituximab combination in unfit patients with CLL.

SECONDARY OUTCOMES:
Number of patients in complete response (CR) or partial response (OR) | At the end of induction therapy, that is, 7 months from treatment start
  Rate of Overall Response Rate (ORR) measured in terms of number of patients in CR/PR at the end of induction therapy.
Number of patients in CR | At the end of induction therapy, that is, at 7 months from treatment start
  Rate of Complete Responses (CR) measured in terms of number of patients in CR at the end of induction therapy.
Number of negative minimal residual disease CRs | At the end of induction therapy, that is, at 7 months from treatment start
  Minimal Residual Disease (MRD) in terms of rate of MRD-negative CRs at the end of induction therapy.
Number of days from treatment discontinuation to new treatment restart. | At the end of the study, that is, 90 months from treatment start
  Time To Next Treatment (TTNT) after treatment discontinuation.
Number of patients in event-free survival | At 36 months from treatment start
  event-Free Survival (PFS) at 36 months.
Number of patients in overall survival (OS) | At 36 months from treatment start
  Overall Survival (OS) at 36 months.
Number of patients in which there is a hematological improvement | At the end of the study, that is, at 90 months from treatment start
  Rate of hematological improvement in patients with baseline anemia, neutropenia and thrombocytopenia defined by hemoglobin >11 g/dL or increase ≥50% over baseline, granulocyte >1500 mm3 or platelet count >100,000/mm3, respectively.
Number of patients with improvement in the immunoglobulin levels | At 90 months from treatment start
  Rate of patients with improvement in the immunoglobulin levels.
Number of adverse events and serious adverse events | At 90 months from study start
Number of patients requiring hospitalization | At 90 months from study entry
  Rate of patients requiring hospitalization, emergency department visits, blood product transfusions and use of hematopoietic growth factors.
Number of patients in which clinical and biological features can be linked | At 90 months from study entry
  Rate of ORR, CR, PFS, EFS, TTNT and OS according to clinical and biologic variables: age, size of nodes, CIRS score, stage, ß2-microglobulin, lymphocyte count, stage, CD38, CD49d, ZAP-70, IGVH mutation status, FISH profile (11q del; 17p del; trisomy 12; 13q del; no aberrations) and mutations of TP53, NOTCH1, SF3B1 and BIRC3.
Number of leukemic subpopulations | At 90 months from start
  Proportion of leukemic and of normal lymphocyte subpopulations, including evaluation of cytokine receptors/adhesion molecules on peripheral blood lymphocytes at week +2 from the start of treatment.
Number of patients with RS identified by FDG-PET/CT | At 90 months from study start
  Rate of cases of patients with RS or SM identified by FDG-PET/CT

CONTACTS AND LOCATIONS:
Overall Officials: Francesca Mauro, Principal Investigator — Policlinico Umberto I di Roma
Locations (36):
- Italy (36):
  - S.O.C. di Ematologia - Azienda Ospedaliera - SS. Antonio e Biagio e Cesare Arrigo, Alessandria
  - U.O.C. Ematologia e Terapia Cellulare - Ospedale "C. e G. Mazzoni" di Ascoli Piceno, Ascoli Piceno
  - S.O.C. di Medicina Interna B - Ospedale - Cardinal Massaia di Asti, Asti
  - UO Ematologia con trapianto-Università degli Studi di Bari Aldo Moro, Bari
  - Istituto di Ematologia "Lorenzo e A. Seragnoli" - Università degli Studi di Bologna - Policlinico S. Orsola - Malpighi, Bologna
  - ASL N.8 - Ospedale "A. Businco" - Struttura Complessa di Ematologia e CTMO, Cagliari
  - U.O.C. di Onco-Ematologia - Centro di Ricerca e Formazione ad Alta tecnologia nelle Scienze Biomediche, Campobasso
  - Unità di Onco-Ematologia - Azienda Ospedaliera - Garibaldi, Catania
  - Azienda Ospedaliera Pugliese Ciaccio - Presidio Ospedaliero A.Pugliese - Unità Operativa di Ematologia, Catanzaro
  - Azienda Ospedaliero Universitaria Arcispedale Sant'Anna Dipartimento di Scienze Mediche Sezione di Ematologia e Fisiopatologia dell'Emostasi, Cona
  - U.O. Ematologia - P.O. Annunziata - A.O. di Cosenza, Cosenza
  - Struttura Complessa di Ematologia Ospedali Riuniti Foggia - Azienda Ospedaliero-Universitaria, Foggia
  - IRCCS_AOU San Martino-IST-Ematologia 1-Monoblocco 11°piano- lato ponente, Genova
  - ASL Le/1 P.O. Vito Fazzi - U.O. di Ematologia ed UTIE, Lecce
  - Istituto Scientifico Romagnoli per lo Studio e la Cura dei Tumori- IRST, Meldola
  - Azienda Ospedaliera Universitaria - Policlinico G. Martino Dipartimento di Medicina Interna - U.O. Messina, Messina
  - Divisione di Ematologia - Azienda Ospedaliera Ospedali Riuniti "Papardo Piemonte", Messina
  - Ospedale Niguarda " Ca Granda" - SC Ematologia Blocco SUD, Ponti Est, Scala E, 4° piano, Milan
  - UO Ematologia - AOU Policlinico di Modena, Modena
  - .C.D.U. Ematologia - DIMECS e Dipartimento Oncologico - Università del Piemonte Orientale Amedeo Avogadro Gianluca Gaidano S.C.D.U. Ematologia - DIMECS e Dipartimento Oncologico - Università del Piemonte Orientale Amedeo Avogadro Novara Davide Rossi S, Novara
  - Università degli Studi di Padova - Ematologia ed Immunologia Clinica, Padua
  - U.O. di Oncoematologia di Nocera Inferiore-plesso ospedaliero "A. Tortora" di Pagani del DEA Nocera-Pagani, Pagani
  - Cattedra di Ematologia CTMO Università degli Studi di Parma, Parma
  - S.C. Ematologia - Fondazione IRCCS Policlinico S. Matteo, Pavia
  - Sezione di Ematologia ed Immunologia Clinica - Ospedale S.Maria della Misericordia, Perugia
  - U.O. Ematologia Clinica - Azienda USL di Pescara, Pescara
  - Dipartimento Oncologico - Ospedale S.Maria delle Croci, Ravenna
  - Dipartimento Emato-Oncologia A.O."Bianchi-Melacrino-Morelli", Reggio Calabria
  - Unità Operativa Complessa di Ematologia - Arcispedale S. Maria Nuova, Reggio Emilia
  - Ospedale "Infermi", Rimini
  - Dipartimento di Biotecnologie Cellulari ed Ematologia - Università degli Studi "Sapienza" di Roma, Roma
  - Università Cattolica del Sacro Cuore - Policlinico A. Gemelli, Roma
  - U.O.C. Ematologia e Trapianti - A.O. Senese - Policlinico " Le Scotte", Siena
  - A.O. Santa Maria - Terni S.C Oncoematologia, Terni
  - Dipartimento di Oncologia ed Ematologia S.C. Ematologia 2 A.O. Città della Salute e della Scienza di Torino San Giovanni Battista, Torino
  - Divisione di Ematologia dell' Università degli Studi di Torino - "Città della Salute e della Scienza di Torino", Torino

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Peragine N, De Propris MS, Intoppa S, Milani ML, Mauro FR, Cuneo A, Rigolin GM, Del Giudice I, Foa R, Guarini A. Early CD49d downmodulation in chronic lymphocytic leukemia patients treated front-line with ibrutinib plus rituximab predicts long-term response. Leuk Lymphoma. 2022 Dec;63(12):2982-2986. doi: 10.1080/10428194.2022.2105324. Epub 2022 Aug 1. No abstract available. PMID 35913400